CLINICAL TRIAL: NCT00542100
Title: PCMRI - an MRI/TRUS System for the Evaluation of the Prostate
Acronym: PCMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TopSpin Medical (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PCL-2-001
Record Dates: First submitted 2007-10-07; First posted 2007-10-10 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: PCMRI
- 2 (Experimental)
  Interventions: Device: PCMRI

INTERVENTIONS:
Device: PCMRI

SUMMARY:
The aim of the clinical study is to evaluate the convenience and efficacy of the PCMRI in the assessment of the prostate in humans.

The study cohort will include 50 patients and is designed to be non-comparative to other diagnostic methods.

DETAILED DESCRIPTION:
Prostate cancer (PC) is the most common male malignancy in the western world. In the U.S. there are approximately 230,000 new diagnoses annually. Each year, 40,000 men with established disease die from PC.

Early detection is possible using prostate specific antigen (PSA) and/or DRE, followed by biopsy if PC is suspected. Biopsy is generally carried out under transrectal ultrasound (TRUS) guidance through the rectum wall. Typically, 6-13 samples from different areas of the prostate are taken in order to cover the entire gland area. Since TRUS cannot accurately detect PC, prostate biopsies, to date, are in fact random biopsies. Furthermore, PSA may be elevated, in patients without PC, leading to as many as 75% of patients undergoing unnecessary TRUS guided biopsy [1,2].

The need for accurate preoperative evaluation of PC, as well as early detection of the tumor has lead to numerous applications of Magnetic Resonance Imaging (MRI) of the prostate.1 The sensitivity and specificity of whole body MRI with pelvic phased-array coils is as low as ~70%. Improved sensitivity is obtained using an endorectal coil where efficacies of ~85% are reported due to the improved signal to noise ratio (SNR) of such coils.2

One of the major limitations of conventional MRI scanners is their cost and limited availability. A portable, hand-held MR scanner capable of detecting PC is thus, of interest. TopSpin has developed a novel MRI based system for prostate imaging in Urology. The primary use of the prostate MRI probe will be diagnosis, staging and guidance of minimally invasive therapy for PC.

The system consists of a miniaturized transrectal MRI probe, incorporating all magnetic field sources and coils. The MRI probe is integrated with and used in conjunction with a TRUS system. The TRUS probe provides prostate gross anatomy and allows the Urologist to select the cross-section(s) of interest within the prostate. The MRI probe provides MRI images of the selected cross-section(s) with improved tissue characterization that enable localizing tumors within the prostate. Fusion of both images has promise of significantly improving the ability to direct biopsies to regions of a much higher likelihood for being malignant. In addition, the system is capable of guiding local treatment such as Cryotherapy or Brachytherapy.

The integrated MRI-TRUS system resembles a state-of-the-art, high-end ultrasound system. The MR-TRUS probe is connected to a cart based console, which houses the electronics hardware required for both MR and ultrasound activation. An investigational device will be manufactured, handled, and stored in accordance with applicable good manufacturing practice (GMP). It will be used in accordance with the approved protocol. Procedures that assure the quality of every aspect of the trial will be implemented.

ELIGIBILITY:
Inclusion criteria for trial group:

* Age between 45 and 80 years old.
* Presumably Stage 2 and higher prostate carcinoma as determined by the PI.
* At least 6 weeks after the last biopsy session.
* Prior to any PC treatment. for control group:
* Age between 25 and 35 years old.
* No family history of PC.
* No lower urinary tract symptoms. Exclusion criteria for both groups:
* History of hemorrhoids.
* History of prostetitis

Ages: 25 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-11; Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the PCMRI system in PC detection | one year
Safety of the PCMRI system in PC detection | one year

SECONDARY OUTCOMES:
Patient comfort | one year
Compliance | one year
Ease of use | one year
Length of the test procedure | one year

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Cytron, MD., Principal Investigator — Barzilai Medical Center, Ashkelon, Israel